CLINICAL TRIAL: NCT00568412
Title: A Multicenter, Randomized, Double-blind Clinical Study to Examine the Efficacy and Safety of Zarzenda in Comparison to Elidel in the Management of Mild to Moderate Atopic Dermatitis in Children and Adolescents
Brief Title: A Clinical Study in Children and Adolescents With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1401920
Record Dates: First submitted 2007-12-03; First posted 2007-12-06 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Mild to Moderate Atopic Dermatitis
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Zarzenda applied topically twice daily for three weeks
  Interventions: Device: Zarzenda
- 2 (Active Comparator): Elidel 1% cream, applied topically twice daily for three weeks
  Interventions: Drug: Elidel

INTERVENTIONS:
Device: Zarzenda — Topical cream, applied twice daily for three weeks
  Arms: 1
Drug: Elidel — 1% cream, applied topically twice daily for three weeks
  Arms: 2

SUMMARY:
To show therapeutic efficacy of Zarzenda cream compared to Elidel cream in children and adolescents with mild to moderate atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* male and female children and adolescents (aged 2 - 17)
* mild to moderate atopic dermatitis
* patients in whom a treatment with topical corticosteroids in not recommended or possible
* wash out periods to be observed

Exclusion Criteria:

* known allergy to one of the two treatments
* known immunodeficiency
* known hepatic or renal insufficiency
* acute skin infections

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment | End of study compared to baseline

SECONDARY OUTCOMES:
EASI | End of study compared to baseline
Affected body surface area | End of study compared to baseline
Patient's assessment of itch, quality of sleep, and global assessment | End of study compared to baseline
Children's Dermatological Life Quality Index | End of study compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Klinik und Poliklinik fuer Dermatologie, Universtitaetsklinikum, Bonn, Germany